CLINICAL TRIAL: NCT05954117
Title: Effect of Chemotherapy on Metabolic Flexibility in the Context of Cachexia in Cancers of the Esophagus and Gastroesophageal Junction
Brief Title: Chemotherapy in the Context of Esophageal and Gastroesophageal Junction Cancer Cachexia
Acronym: CHIFMEOE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other); Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AOI 2022 RICHARD; 2023-A00582-43 (Other: ANSM)
Record Dates: First submitted 2023-06-16; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Adenocarcinoma
Keywords: Mitochondria; Oxygraphy; Adipose Tissue; Gastroesophageal adenocarcinoma; Energy expenditure
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

STUDY DESIGN:
Intervention Model Description: patient undergoing surgery for esophageal adenocarcinoma or for gastroesophageal adenocarcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): patients with esophageal or gastroesophageal adenocarcinoma included to evaluate the energy expenditure before and after chemotherapy and evaluate parameters of cachexia
  Interventions: Procedure: Adipose tissue biopsies

INTERVENTIONS:
Procedure: Adipose tissue biopsies — During the 2 surgical time, when patient is under general anesthesia, two adipose tissue biopsies of 20cc each (one from abdominal subcutaneous adipose tissue and one from omental adipose tissue) are taken and characterize by oxygraphy (respirometry).
  Before the 2 surgical times (before and after chemotherapy) patients will have evaluation of the muscle strength, cachexia (by scan analysis), energy expenditure, anthropometric criteria and biochemical inflammatory.

SUMMARY:
Cachexia is a syndrome frequently associated with digestive cancers and more particularly with esophageal and gastroesophageal adenocarcinoma. Its pathophysiology remains poorly understood, multi-factorial, but strongly correlated to the prognosis of patients. It's a consequence of the imbalance of energy balance linked to tumoral process, to dysphagia and to anorexia, frequently present in these cancers. At the center of this imbalance, adipose tissue plays a major role. Recent studies showing that the mobilization of lipid substrates and the hypermetabolism of adipocytes are involving in its development, even before loss of muscle. As part of the management, neoadjuvant chemotherapy is usually administered with the main objective to reduce tumor extension and dissemination through actions on DNA and mitosis. These treatments will also alter the mitochondrial function of cells in other tissues, probably including that of adipocytes. A paradoxical effect on the cachectic process could thus be envisaged, as a decrease in mitochondrial activity and associated hypermetabolism, and therefore a preservation of fat mass, and by extension of muscle mass.

Primary endpoint: identify the adipocyte factors involved in the energy imbalance associated with the cachectic process in patients managed for esophageal or gastroesophageal adenocarcinoma.

Secondary endpoint: compare the results obtained before and after chemotherapy treatment according to the cachectic state and the anatomical location of the adipose sample (subcutaneous versus visceral) to evaluate the resting energy expenditure.

DETAILED DESCRIPTION:
Two operative steps, separated by neoadjuvant chemotherapy, are classically planned in the management of esophageal and gastroesophageal adenocarcinoma: an exploratory laparoscopy as part of the disease extension assessment and the tumor resection surgery (esophagectomy). During these operations, the surgeon will perform a subcutaneous fat biopsy at the surgical approach and a visceral fat biopsy at the epiploic level. A portion of the samples will be immediately analyzed by high-resolution oxygraphy to evaluate the mitochondrial metabolism of the adipocytes. The rest of biopsies will be frozen for further biological analysis (enzymology, Western-blot, RT-qPCR) or embedded in paraffin for histological analysis (morphometry, inflammation, metabolism). Serum will also be recovered with the biopsies for specific biological analysis (inflammatory and lipid status).

In days preceding the interventions, in addition to the usual management, will be performed: an evaluation of the energy expenditure by indirect calorimetry, an evaluation of the body composition by Dual Energy X-ray Absorptiometry (DEXA), physical tests to evaluate sarcopenia and cachexia, nutritional and quality of life questionnaires, and a medical examination with a dietetic consultation.

ELIGIBILITY:
Inclusion Criteria:

* Male Patients
* Patients aged over 18
* Patients eligible for neoadjuvant FLOT chemotherapy (5-fluorouracil, oxaliplatin, docetaxel);
* Patients with a resealable adenocarcinoma of esophageal or gastroesophageal
* Patients able to give informed consent.
* Patients affiliated to a Health Care insurance

Exclusion Criteria:

* Unresectable or metastatic esophageal or gastroesophageal adenocarcinoma;
* Another tumor histology than adenocarcinoma.
* Patients not eligible for neoadjuvant FLOT chemotherapy and/or for surgery
* Patients under guardianship, curators or deprived of liberty;
* Refusal to participate;
* Patients already participating in another interventional study of pharmacological, nutritional and/or rehabilitation study;
* Patients in a period of exclusion from another research protocol.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of mitochondrial respiration on adipose tissue by oxygraphy | 6 week
  Evaluation of mitochondrial respiration on adipose tissue before and after chemotherapy Mitochondrial respiration measurements in oxydo-phosphorylated conditions. For each patient measurements using ADP and carbohydrate or lipid substrates of the respiratory chain complexes for both the subcutaneous and the visceral tissue.

SECONDARY OUTCOMES:
Evaluation of sarcopenia (SARC-F : sarcopenia scoring) | 1 week
  level of sarcopenia between 0 to 12 including 5 questions
anthropometric data | 1 week
  BMI will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, Principal Investigator — Ruddy.Richard@Uca.Fr
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bacoeur-Ouzillou O, Guerrier L, Touron J, Pinel A, Pereira B, Meunier N, Gillet B, Pezet D, Cassagnes L, Malpuech-Brugere C, Richard R, Gagniere J. Chemotherapy effects on mitochondrial function in adipose tissue in oesophageal and gastroesophageal junction adenocarcinomas with or without associated cachexia: protocol for a prospective, comparative observational study (ChiFMeOE). BMJ Open. 2024 Oct 23;14(10):e086686. doi: 10.1136/bmjopen-2024-086686. PMID 39448207